CLINICAL TRIAL: NCT02336087
Title: A Pilot Study of Gemcitabine, Abraxane, Metformin and a Standardized Dietary Supplement (DS) in Patients With Unresectable Pancreatic Cancer
Brief Title: Gemcitabine Hydrochloride, Paclitaxel Albumin-Stabilized Nanoparticle Formulation, Metformin Hydrochloride, and a Standardized Dietary Supplement in Treating Patients With Pancreatic Cancer That Cannot be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14122; NCI-2014-02612 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14122 (Other: City of Hope Medical Center)
Record Dates: First submitted 2015-01-06; First posted 2015-01-12 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Adenocarcinoma; Unresectable Pancreatic Carcinoma; Stage III Pancreatic Cancer AJCC v6 and v7; Stage IV Pancreatic Cancer AJCC v6 and v7
MeSH Terms: interventions — Gemcitabine; Taxes; Albumin-Bound Paclitaxel; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (gemcitabine, Abraxane, metformin, DS) (Experimental): Patients receive gemcitabine hydrochloride and paclitaxel albumin-stabilized nanoparticle formulation IV on days 1, 8, and 15. Patients also receive metformin hydrochloride PO BID starting day -6 and dietary supplement PO BID starting day -3. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine Hydrochloride; Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation; Drug: Metformin Hydrochloride; Dietary Supplement: Therapeutic Dietary Intervention; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdC; dFdCyd
Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation — Given IV
  Other Names: ABI 007; ABI-007; Abraxane
Drug: Metformin Hydrochloride — Given PO
  Other Names: Glucophage; Metformin HCl
Dietary Supplement: Therapeutic Dietary Intervention — Given PO
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot phase I trial studies the side effects of gemcitabine hydrochloride, nab-paclitaxel, metformin hydrochloride, and a standardized dietary supplement in treating patients with pancreatic cancer that cannot be removed by surgery. Drugs used in chemotherapy, such as gemcitabine hydrochloride and paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Metformin hydrochloride, used for diabetes, may also help kill cancer cells. Dietary supplements (curcumin, vitamin D, vitamin K2, vitamin K1, B-6, high selenium broccoli sprouts, epigallocatechin gallate, L-carnitine, garlic extract, genistein, zinc amino chelate, mixed toxopherols, ascorbic acid, D-limonene) can block different targets in the cancer cell simultaneously and may slow down cancer growth. Giving gemcitabine hydrochloride, paclitaxel albumin-stabilized nanoparticle formulation, and metformin hydrochloride with a dietary supplement may work better in treating patients with pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the compliance, toxicity and feasibility of administering gemcitabine hydrochloride (gemcitabine), nab-paclitaxel (abraxane), metformin hydrochloride (metformin), and the dietary supplement (DS).

SECONDARY OBJECTIVES:

I. To assess the response rate associated with this combination therapy in pancreatic cancer patients.

II. To assess the progression-free survival and overall survival of all patients who start protocol therapy, and describe the outcomes based on measures of compliance during the lead-in week, and compliance with supplement during chemotherapy.

III. To collect and analyze peripheral blood and pre-treatment biopsy samples for an exploratory analysis of biological correlatives.

IV. To assess quality of life utilizing the Functional Assessment of Cancer Therapy-General (FACT-G) questionnaire.

OUTLINE:

Patients receive gemcitabine hydrochloride and paclitaxel albumin-stabilized nanoparticle formulation intravenously (IV) on days 1, 8, and 15. Patients also receive metformin hydrochloride orally (PO) twice daily (BID) starting day -6 and dietary supplement PO BID starting day -3. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologic diagnosis of pancreatic adenocarcinoma
* Patient must have unresectable disease
* Patients must not have received prior chemotherapy except for the following circumstances; gemcitabine and capecitabine chemotherapy given in the adjuvant setting is allowed if the recurrence is greater than 6 months from the completion of chemotherapy; radiation sensitizing doses of 5-fluororuracil or capecitabine are allowed as part of adjuvant treatment and recurrence must be documented greater than 6 months from the completion of adjuvant therapy
* Computed tomography (CT) or magnetic resonance imaging (MRI) scan must be obtained within 4 weeks prior to study entry
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Absolute neutrophil count > 1,500/mcl
* Platelet count > 100,000/mcl
* Creatinine < 1.4 mg/dl and/or a measured creatinine clearance > 60 cc/min
* Bilirubin < 1.4 mg/dl
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) no greater than 3.0 times the upper limit of normal
* Patients currently being treated for severe infections or who are recovering from major surgery or other intercurrent illnesses are ineligible until recovery is deemed complete by the investigator
* Patients must not be pregnant or nursing; women and men of reproductive potential must have agreed to use an effective contraceptive method
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* Patients must be able to swallow pills and must not have malabsorption problems or ongoing nausea and vomiting that would affect oral treatment
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* Patients currently taking metformin will be eligible
* Patients allergic to eggs are not eligible
* Patients taking additional dietary/herbal supplements (excluding Senekot) outside of this protocol and refusing to stop are not eligible
* Patients requiring warfarin are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2020-10-04 (Actual); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the combination of gemcitabine hydrochloride, paclitaxel albumin-stabilized nanoparticle formulation, metformin hydrochloride, and a dietary supplement | Up to 24 months
  Feasibility is defined at 1 or fewer patients experiencing a dose limiting toxicity within the first 6 patients.
Compliance of the combination of gemcitabine hydrochloride, paclitaxel albumin-stabilized nanoparticle formulation, metformin hydrochloride, and a dietary supplement (percent of patients who are fully compliant) | Up to 24 months
  The percent of patients who are fully compliant in the first week will be estimated with a 95% confidence interval. The compliance will be measured similarly for each course prior to study treatment discontinuation. The impact of less than full compliance (both during the lead-in period and during chemotherapy) on the biomarkers and outcome, and qualitatively study patient reasons and specific supplement patterns related to non-compliance will be explored.
Toxicity of the combination of gemcitabine hydrochloride, paclitaxel albumin-stabilized nanoparticle formulation, metformin hydrochloride, and a dietary supplement (National Cancer Institute Common Terminology for Adverse Events criteria version 4) | Up to 24 months
  Summarized using the National Cancer Institute Common Terminology for Adverse Events criteria version 4. Tables will summarize the highest grade per patient that is possibly related to treatment, and the number of patients requiring dose modifications will also be presented.

SECONDARY OUTCOMES:
Progression-free survival | Up to 24 months
  Evaluated using the Kaplan-Meier methods.
Overall survival | Up to 24 months
  Evaluated using the Kaplan-Meier methods.
Time to treatment failure | Up to 24 months
  Evaluated using the Kaplan-Meier methods.

OTHER OUTCOMES:
Analysis of biological correlates (Peripheral blood will be evaluated) | Up to 24 months
  Peripheral blood will be evaluated. Standard descriptive methods will be used to summarize the baseline levels and the changes from baseline (i.e. after treatment) in order to examine whether observed patterns are consistent with hypothesized patterns.
Quality of life, assessed using the FACT-G questionnaire | Up to 24 months
  Standard descriptive methods will be used to summarize the baseline levels and the changes from baseline (i.e. after treatment) in order to examine whether observed patterns are consistent with hypothesized patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chung, Principal Investigator — City of Hope Medical Center
Locations (4):
- United States (4):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Rancho Cucamonga, Rancho Cucamonga, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope West Covina, West Covina, California